CLINICAL TRIAL: NCT04290663
Title: Multicentric Phase III Trial Comparing Two Strategies in Intermediate-risk Differentiated Thyroid Cancer Patients: Systematic Radioiodine Administration Versus Decision of Radioiodine Treatment Guided by a Post-operative Work-up Based on Serum Tg Values and Diagnostic RAI Scintigraphy
Brief Title: Systematic Radioiodine Administration Versus Decision of Radioiodine Treatment Guided by a Post-operative Work-up
Acronym: INTERMEDIATE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: French cancer Institute INCa (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-002968-27
Record Dates: First submitted 2020-02-20; First posted 2020-03-02 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Cancer; Intermediate Risk
Keywords: radioiodine; I131
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAI group (Active Comparator)
  Interventions: Drug: Systematic RAI-treatment
- GUIDED FOLLOW-UP group (Experimental)
  Interventions: Other: Decision of RAI-treatment guided by a post-operative assessment

INTERVENTIONS:
Drug: Systematic RAI-treatment — Administration of 3.7 GBq (100 mCi) or 1,1 GBq (30 mCi) of I131 at the choice of the investigator after rhTSH-stimulation
  Arms: RAI group
Other: Decision of RAI-treatment guided by a post-operative assessment — The decision-making for the administration of an adapted RAI-treatment will be taken according to the following criteria:
  * No RAI treatment if Tg/LT4 ≤1 ng/mL and rhTSH-sTg ≤10 ng/mL and normal diagnostic RAI-scintigraphy
  * 1.1 GBq after rhTSH if Tg/LT4>1 ng/mL or rhTSH-sTg>10 ng/mL and normal diagnostic RAI-scintigraphy.
  * 3.7 GBq after rhTSH if metastatic lymph-node(s) detected on diagnostic RAI-scintigraphy without distant metastasis
  * 3.7 GBq after hormone withdrawal if distant metastasis detected on diagnostic RAI-scintigraphy or on the hybrid CT scan of the SPECT-CT acquisition
  Arms: GUIDED FOLLOW-UP group

SUMMARY:
This trial is comparing two strategies in intermediate-risk differentiated thyroid cancer patients: Systematic radioiodine administration versus decision of radioiodine treatment guided by a post-operative work-up based on serum Tg values and diagnostic RAI scintigraphy

ELIGIBILITY:
Inclusion Criteria:

* Subgroup of patients with differentiated thyroid cancer and intermediate-risk defined as follows according to TNM 2017:

  * Papillary thyroid cancer (PTC) without aggressive subtype, follicular thyroid cancer (FTC) (with < 4 foci of vascular invasion) or Hürthle cell carcinoma (HCC)
  * T1b or T2 with minimal extra-thyroid extension into the perithyroidal soft tissues and/or pN1 with largest nodal dimension between 2 and 10 mm, without extra-capsular invasion and with a number of metastatic nodes ≤ 10
  * T1aN1 with largest nodal dimension between 2 and 10 mm, without extra-capsular invasion and with a number of metastatic nodes ≤ 10
* Patient treated by total thyroidectomy with macroscopically complete tumor resection (R0 or R1) ± neck dissection
* Total thyroidectomy performed within 6 to 14 10 weeks before randomization
* Patient with or without anti-thyroglobulin antibodies (TgAb)
* No known distant metastases
* Normal post-operative neck ultrasound (US) or if doubtful US, negative cytology and normal Tg value (<10 ng/ml) in FNA washout fluid
* Post-operative LT4 treatment initiated at least 6 weeks before randomization
* Performance Status 0 or 1
* Patients aged 18 years or older
* Signed informed consent form
* Patient who agrees to be followed annually during 5 years
* Patient affiliated to the French social security system

Exclusion Criteria:

* • Patients with:

  * medullary or anaplastic thyroid cancer
  * or poorly differentiated carcinoma
  * or well differentiated FTC with at least more than 4 foci of vascular invasion
  * or PTC with aggressive variants (tall cell or columnar cell carcinoma, diffuse sclerosing papillary, hobnail variant)
  * NIFTP (Noninvasive follicular thyroid neoplasm with papillary-like nuclear features)

    • Low-risk or high-risk DTC patients according to ATA 2015, and intermediate-risk patients with extra-thyroid extension into the perithyroidal muscles (pT3b according to pTNM 2017), and/or pN1 with nodal largest dimension >10 mm or with extra-capsular invasion or more than 10 metastatic nodes. This excludes the following patients:
  * All pT1a, pT3 or pT4
  * pT1aN0/x with or without minimal extra-thyroid extension
  * pT1bN0/x, pT2N0/Nx without minimal extra-thyroid extension
  * pT1aN1 or pT1bN1 or pT2N1 without extra-thyroid extension and with nodal largest dimension <2mm
  * pT1aN1 or pT1bN1 or pT2N1 without extra-thyroid extension and with nodal largest dimension >10mm
  * pT2N0/Nx without extra-thyroid extension
  * pT2N1 without extra-thyroid extension and with nodal largest dimension <2mm
  * pT2N1 without extra-thyroid extension and with nodal largest dimension >10mm
  * Surgery considered as macroscopically incomplete (R2)

    * Patients who have undergone lobectomy only
    * Post-operative neck US with metastatic lymph-nodes confirmed by cytology or by increased Tg (>10 ng/ml) in FNA washout fluid
    * Drugs affecting thyroid function including iodinated contrast agents in the 6 weeks prior to randomization. Amiodarone should have been stopped at least 1 year before randomization.
    * Previous RAI treatment for thyroid cancer
    * Pregnant or lactating women
    * Any associated geographical, social or psychopathological condition that could compromise the patient's ability to participate in the study
    * Patient deprived of liberty or placed under the authority of a tutor
    * History of malignancy in the past 3 years, except skin cancer excluding melanoma, carcinoma in situ of the cervix. Any other solid tumor or lymphoma (without bone marrow involvement) must have been treated and not have shown signs of recurrence for at least 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2031-02 (Estimated); Study Completion 2033-02 (Estimated)

PRIMARY OUTCOMES:
the rate of patients with excellent tumoral response | 36 months after randomization
  normal neck ultrasonography and Tg/LT4 <0.2 ng/mL and absence of TgAb and if performed, no abnormalities on other imaging modalities

SECONDARY OUTCOMES:
Patient's quality-of-life | During I131 treatment and at 1 and 3 years
  Comparison of the scores on SF-36 (score between 0 and 100) between 2 arms
Salivary, nasal and lachrymal toxicities | During I131 treatment and at 1,2,3 and 5 years
  Comparison of the intensity of salivary, nasal and lachrymal toxicities between 2 arms
Management cost | through study completion, an average of 5 years
  Costs of all medical exams and transportation related to the care within 5 years post-randomization in both groups
Patient's anxiety | During I131 treatment and at 1 and 3 years
  Comparison of the scores on STAI questionnaire (score between 20 and 80) between 2 arms

CONTACTS AND LOCATIONS:
Locations (29):
- France (29):
  - CHU Pointe à pitre, Pointe à Pitre, Guadeloupe
  - Chu Angers, Angers
  - Institu de Cancérologie de l'Ouest - Site Angers, Angers
  - Bergonié, Bordeaux
  - Hôpital saint-André, Bordeaux
  - Chu Brest, Brest
  - Centre Francois Baclesse, Caen
  - Centre Hospitalier Métropôle Savoie, Chambéry
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges-François Leclerc, Dijon
  - Chu Martinique, Fort de France
  - Chu Grenoble, Grenoble
  - Chru Lille, Lille
  - Centre Léon Bérard, Lyon
  - Hospices Civils de Lyon, Lyon
  - CHU Timone, Marseille
  - Chu Nancy, Nancy
  - Chu Nantes, Nantes
  - Centre Antoine Lacassagne -, Nice
  - Chu Nimes, Nîmes
  - AP-HP Pitié Salpétrière, Paris
  - Centre Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Institut CURIE, site Réné Huguenin, Saint-Cloud
  - Institu de Cancérologie de l'Ouest - Site St Herblain, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - CHU TOULOUSE, Hôpital Larrey, Toulouse
  - IUCT Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No